CLINICAL TRIAL: NCT03821766
Title: Do Abnormal Hemodynamic Features Generate Relevant Reactions and Vibrations at the Skin Level When Recorded by Micro Accelerometers
Brief Title: Haemodynamic Abnormalities Recorded With Cardiac Catheterization Along With Body's Surface Micro-accelerometers (KT-KCG)
Acronym: KT-KCG
Status: Withdrawn | Type: Observational
Why Stopped: Technical failure
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2018/479
Record Dates: First submitted 2019-01-11; First posted 2019-01-30 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-08

CONDITIONS: Heart Failure; Pulmonary Hypertension
Keywords: Intracavitary pressure; Ballistocardiography; Seismocardiography; Microaccelerations; Kinetic energy
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — Ballistocardiography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Heart failure: Patients suffering from heart failure regardless to the etiology will undergo cardiac catheterization according to their medical condition. the SCG and BCG signals will be recorded along with the intracavitary pressure profiles detected invasively with the cardiac catheterization.
  Interventions: Device: Ballistocardiography and seismocardiography

INTERVENTIONS:
Device: Ballistocardiography and seismocardiography — SCG and BCG signals will be recorded by the mean of an unobtrusive and friendly device consisting of two houses, the first one placed on the sternum and the second one place on the lumbar region near the subject's center of mass. The signal will be transferred to a tablet by Bluetooth and tracings will be analysed automatically with Matlab. The SCG+BCG signals are synchronized to the intracardiac pressure tracings in order to allow a comparative interpretation between the two tracings.

SUMMARY:
The ballistocardiography (BCG) and the seismocardiography (SCG) are old techniques recording the vibrations at the skin level generated by the acceleration and displacement of the blood and cardiac mass at each cardiac contraction. The former records the acceleration near the subject's center of mass, the latter at the local chest wall. So far, the unclear physiological origin of those acceleration signals has led to important ambiguities in their scientific and clinical interpretation. Therefore, several ongoing studies would aim to highlight the physiological genesis of those acceleration-induced signals.

Indeed, the main objective of this study is to correlate the BCG and SCG signals recorded at the body surface with several haemodynamic parameters recorded invasively during a cardiac catheterisation, pulmonary pressure, wedge pressure, cardiac output to cite a few.

DETAILED DESCRIPTION:
Patients suffering from severe heart failure regardless of the etiology will undergo a cardiac catheterization as required by their medical condition.

The SCG and BCG signals will be recorded simultaneously to the catheterization by the mean of an unintrusive and friendly device consisting of two houses, the first one placed on sternum and the second one in the lumbar column. The device will record a continuous tracing synchronized with the intracavitary pressure profiles recorded during the invasive procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 y.o. to 80 y.o.
* Heart failure

Exclusion Criteria:

* Left ventricle assistance device
* Refused participation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from heart failure and undergoing a planned cardiac catheterization as required by their medical condition will be asked to participate to the study.
  The inclusion criteria include heart failure regardless of its etiology. Patients with a left ventricle assistance device will not be enrolled because the high-frequency accelerations generated by the mechanical device and transmitted to the skin level will likely hamper the ballisto- and seismocardiographic signal.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Micro-accelerations recorded at the body's surface | 6 months
  Analysis of heart-induced velocities (m/s) by the means of micro-accelerometers and secondary computation of the kinetic energy (KE= 1/2 mv²) recorded with the seismocardiography and ballistocardiography at the skin level during cardiac catheterization.

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2019-01-25): https://cdn.clinicaltrials.gov/large-docs/66/NCT03821766/Prot_000.pdf